CLINICAL TRIAL: NCT03113903
Title: Validation of the French Version of the Pain Sensitivity Questionnaire
Acronym: PSQ-F
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Inserm U1107 " Neuro-Dol ", Clermont-Ferrand, France (Unknown); Centre Jean Perrin (Other); Klinikum der Universität München, Deutschland (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: CHU-311; 2016-A02079-42 (Other: 2016-A02079-42)
Record Dates: First submitted 2017-03-20; First posted 2017-04-14 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2018-11

CONDITIONS: Scheduled Surgery; Healthy Volunteers
Keywords: Pain; psychophysics; Nociception; Sensitivity; Senses; Phenotyping; Questionnaire; Anxiety; Depression; Catastrophizing
MeSH Terms: conditions — Pain; Hypersensitivity; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant
Masking Description: open
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- scheduled surgery (Experimental)
  Interventions: Behavioral: Psychophysical exploration
- healthy volunteers (Other)
  Interventions: Behavioral: Psychophysical exploration

INTERVENTIONS:
Behavioral: Psychophysical exploration — Psychophysical exploration (multimodal sensitivity, including pain sensitivity) Electronic von Frey applied on forearm; thermal heat applied on forearm; foot immersion in 2°C cold water; exposure to a one-frequency noise up to uncomfortable loudness ; exposure to a halogen-lamp-generated light up to uncomfortable brightness.

SUMMARY:
The Pain Sensitivity Questionnaire (PSQ) is a tool created in 2009 by Dr. R. Ruscheweyh in Germany. It aims at identifying the natural sensitivity to pain, through a set of 17 simple questions. These questions simulate daily life situations likely to induce pain of various intensities. The internal validity of the tool had been demonstrated both for the original version in German, and then for its English version. The external validity had also been demonstrated by correlation to real nociceptive stimulations applied to healthy volunteers (German version), and to patients before surgery (English version). A French validation of the questionnaire is needed, in order to integrate it in pain research programs in French-speaking countries.

DETAILED DESCRIPTION:
The aim is to validate the French version of the PSQ in a 2-step plan : (i) validity of internal structure, convergent validity and reproducibility, in a sample of patients before scheduled surgery, and (ii) structure and convergent validity against external criterion, in healthy volunteers. A secondary objective is to study the relationship of scores of the PSQ with a scale assessing sensitivity to natural smells, noise and light sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 to 65, currently French-speaking and able to answer questionnaires, undergoing a pre-anesthetic mandatory visit, either for scheduled surgery, or as a follow-up of pregnancy
* healthy volunteers aged 18 to 60, currently French-speaking and able to answer questionnaires, BMI 19 to 30 kg/m2, free from any medication since 7 days before each study session, covered by the French welfare health system. Exclusion criteria are : risk of pregnancy, any medical history or condition likely to impair participation or quality of outcome measurement, any ongoing relevant disease, any cutaneous lesion at nondominant forearm, any ocular, neurological or acoustic contra-indication to the tests, spontaneous tinnitus or disease with hyperacusia, anxiety or depression with score >11 on HAD, addiction to drugs or alcohol abuse, inclusion in a concomitant trial, French legal protection

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2017-04-30 (Actual); Primary Completion 2018-01-23 (Actual); Study Completion 2018-01-23 (Actual)

PRIMARY OUTCOMES:
The psychometric properties of the French version of the PSQ | at day 1
  (acceptability, internal validity, reproducibility, convergent validity and validity of structure against external criteria)

SECONDARY OUTCOMES:
The natural smell sensitivity assessed independently by a home-made questionnaire | at day 1
  one measurement point
The natural noise sensitivity assessed independently by a home-made questionnaire | at day 1
  one measurement point
The natural light sensitivity, assessed independently by a home-made questionnaire | at day 1
  one measurement point

CONTACTS AND LOCATIONS:
Overall Officials: Christian DUALE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Background] Duale C, Bauer U, Storme B, Eljezi V, Ruscheweyh R, Eschalier S, Dubray C, Guiguet-Auclair C. Transcultural adaptation and French validation of the Pain Sensitivity Questionnaire. Can J Anaesth. 2019 Oct;66(10):1202-1212. doi: 10.1007/s12630-019-01377-w. Epub 2019 Apr 24. PMID 31020630
- [Derived] Duale C, Leray V, Giron F, Boulliau S, Macian N, Ruscheweyh R, Dubray C, Giraudet F. The Added Value of Sensitivity to Nonnoxious Stimuli to Predict an Individual's Sensitivity to Pain. Pain Physician. 2021 Sep;24(6):E783-E794. PMID 34554698